CLINICAL TRIAL: NCT01270698
Title: A Phase I Study of IMMU-130 (hMN-14-SN38 Antibody Drug Conjugate) in Patients With Colorectal Cancer.
Brief Title: Study of IMMU-130 in Patients With Relapsed/Refractory Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-IMMU-130-01
Record Dates: First submitted 2011-01-03; First posted 2011-01-05 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2015-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — labetuzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMMU-130 (Experimental)
  Interventions: Drug: IMMU-130

INTERVENTIONS:
Drug: IMMU-130 — IMMU-130 will be administered intravenously every 2 weeks for up to 6 months or longer.
  Other Names: hMN14-SN38

SUMMARY:
This is a Phase I trial to study the safety of IMMU-130. IMMU-130 is composed of a drug attached to an antibody. The drug is the active ingredient in irinotecan which is a common chemotherapy drug used for colorectal cancer. Antibodies are proteins normally made by the immune system. They bind to substances that don't belong in the body to prevent harm to the body. The antibody in this study was designed to bind to a marker located on colorectal cancer tumors. The antibody was originally made from mouse proteins, but was changed in the laboratory to be more like human antibodies. This study will investigate how IMMU-130 acts for the treatment of colorectal cancer. The study is mainly being done to see if IMMU-130 is safe.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, >18 years of age, able to understand and give written informed consent.
* Histologically or cytologically confirmed colorectal adenocarcinoma.
* Stage IV (metastatic) disease.
* Failed at least one prior standard treatment regimen for colorectal cancer
* Adequate performance status (ECOG 0 or 1)
* Expected survival > 6 months.
* CEA plasma levels > 5 ng/mL
* Measurable disease by CT or MRI
* At least 4 weeks beyond major surgery and recovered from all acute toxicities
* At least 2 weeks beyond corticosteroids, except low doses (i.e., 20 mg/day of prednisone or equivalent) to treat nausea or other illness such as rheumatoid arthritis
* Adequate hematology without ongoing transfusional support (hemoglobin > 9 g/dL, ANC > 1,500 per mm3, platelets > 100,000 per mm3)
* Adequate renal and hepatic function (creatinine ≤ 1.5 x IULN, bilirubin ≤ IULN, AST and ALT ≤ 3.0 x IULN or 5 x IULN if know liver metastases).
* Otherwise, all toxicity at study entry <Grade 1 by NCI CTC v4.0.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Women of childbearing potential and fertile men unwilling to use effective contraception during study until conclusion of 12-week post-treatment evaluation period.
* Patient's with Gilbert's disease or known CNS Metastatic disease. However, patients with CNS metastases who are asymptomatic and have completed a course of therapy are eligible for the study provided they are clinically stable for 1 month prior to entry as defined as: (1) no evidence of new enlarging CNS metastasis (2) off steroids or on a stable dose of steroids
* Patients with CEA plasma level > 1000 ng/mL are excluded during dose escalation, but may be included after the MTD is determined
* Patients with active grade 3 anorexia, nausea or vomiting, and/or signs of intestinal obstruction.
* Patients with non-melanoma skin cancer or carcinoma in situ of the cervix are not excluded, but patients with other prior malignancies must have had at least a 3-year disease free interval.
* Patients known to be HIV positive, hepatitis B positive, or hepatitis C positive.
* Known history of unstable angina, MI, or CHF present within 6 months or clinically significant cardiac arrhythmia (other than stable atrial fibrillation) requiring anti-arrhythmia therapy,
* Known history of clinically significant active COPD, or other moderate-to-severe chronic respiratory illness present within 6 months.
* Known autoimmune disease or presence of autoimmune phenomena (except rheumatoid arthritis requiring only low dose maintenance corticosteroids, and other than diabetes, vitiligo, or stable thyroid disease).
* Infection requiring intravenous antibiotic use within 1 week.
* Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety | Safety will be measured routinely during the 6 months of administration and afterwards during follow-up for up to 5 years
  The primary outcome measured will be safety of IMMU-130 administered at different dose levels. Safety will be assessed by reviewing the number of adverse events and overall toxicity.

SECONDARY OUTCOMES:
efficacy | Efficacy will be measured every 8-12 weeks during treatment and every 6 months during the 2nd year and then annually up to 5 years thereafter.
  The secondary objectives are to assess pharmacokinetics and immunogenicity, and to obtain preliminary information on efficacy with this dosing schedule. Efficacy will be assessed using CT scan imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States